CLINICAL TRIAL: NCT05391542
Title: Effectiveness of Tubular Coaxial Nickel-titanium and Copper Nickel-titanium Orthodontic Aligning Archwires: A Randomized Clinical Trial
Brief Title: Effectiveness of Tubular Coaxial Nickel-titanium and Copper Nickel-titanium Orthodontic Aligning Archwires
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Reyam Mohammed Noori, Orthodontics master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 599422
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aligning Archwires

STUDY DESIGN:
Intervention Model Description: The patients will be treated with straight wire appliance using MBT prescription brackets with 0.022-inch slot (Pinnacle®, Ortho Technology, USA). Initially, teeth polishing will be performed with pumice and rubber cup, followed by water rinsing and air drying
  Archwire sequence for each group will be as follows:
  1. Coaxial tubular superelastic nickel-titanium Group (TuNT) (Speed tubular supercable, Speed System™ Orthodontics, Ontario, Canada):
     * 0.016-inch
     * 0.018-inch
  2. Copper-nickel-titanium Group (CuNT) (Damon Optimal-Force Copper Ni-Ti®, Ormco, Glendora, Calif):
     * 0.014-inch
     * 0.018-inch Allocation Concealment: This will be achieved using sequentially numbered, opaque and sealed envelopes which will be numbered according to the study numbers. Each envelope includes the treatment allocation card (group 1 or 2) and the related archwires.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sequence Generation: A computer random generator will be used to develop a simple randomization with an equal allocation ratio (1:1) and without stratification.
  Allocation Concealment: This will be achieved using sequentially numbered, opaque and sealed envelopes which will be numbered according to the study numbers. Each envelope includes the treatment allocation card (group 1 or 2) and the related archwires.
  Blinding As the study will be conducted in different clinics, all data collection and measurement will be completed with the investigator being masked to the allocation groups, though blinding of the operator will not be possible during the archwire placement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaxial tubular superelastic nickel-titanium Group (TuNT) (Experimental): 0.016-inch coaxial tubular superelastic nickel-titanium archwire (TuNT) (Speed tubular supercable, Speed System™ Orthodontics, Ontario, Canada) will be placed in mandibular arch at the day of bonding. Eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks
  Interventions: Other: aligning archwires
- Copper-nickel-titanium Group (CuNT) (Experimental): 0.014-inch Copper-nickel-titanium archwire (CuNT) (Damon Optimal-Force Copper Ni-Ti®, Ormco, Glendora, Calif) will be placed in mandibular arch at the day of bonding. Eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks.
  Interventions: Other: aligning archwires

INTERVENTIONS:
Other: aligning archwires — At the day of bonding, 0.016-inch archwire will be placed for the TuNT group. Eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks. While, for the CuNT group, 0.014-inch archwire will be placed at the day of bonding and eight weeks later it will be replaced by the 0.018-inch archwire for another eight weeks. Archwires will be tied to the bracket by elastomeric modules which will be changed every 4 weeks. A good-quality alginate impression for the lower arch should be taken pre-treatment and after 4, 8, 12 and 16 weeks and a stone study model is obtained. Periapical X-ray for the mandibular central incisors will be taken pre-treatment and after 16 weeks. The participants will be provided by a visual analog scale (0-10) to record their pain perception during the first week after each wire placement.

SUMMARY:
This study will be done to compare the effectiveness of using coaxial tubular superelastic nickel-titanium and copper-nickel-titanium archwires during the initial phase of orthodontic treatment regarding alignment efficiency, pain perception, and root resorption.

DETAILED DESCRIPTION:
This will be a prospective blinded non-stratified randomized clinical trial , parallel group trial with equal randomization (1:1 allocation ratio), different private clinics and general hospitals will allocate patients for this trial. The patients will be initially assessed for eligibility to be included in the study by the investigator. Those who will meet the inclusion criteria will be informed about the nature of the study verbally to take the initial approval for participation. The patients were asked to read the patient information sheet carefully at home and inform the investigator about their decision of participation at the subsequent appointment and to sign consent form sheet in case of agreement.

The patients will be treated using MBT prescription brackets with 0.022-inch slot (Pinnacle®, Ortho Technology, USA). Initially, teeth polishing will be performed with pumice and rubber cup, followed by water rinsing and air drying

All the participants will receive the same treatment. At the day of bonding, the first archwire will be placed for each group. Eight weeks later it will be replaced by the next size archwire for another eight weeks. Archwires will be tied to the bracket using elastomeric ligatures. Any debonding during treatment should be considered an emergency and re-bonded within 24 hours, otherwise the case will be dropout. A good alginate impression for the lower arch should be taken pre-treatment and after 4, 8, 12 and 16 weeks and a stone study model is obtained. Periapical X-ray for the mandibular central incisors will be taken pre-treatment and after 16 weeks. The participants will be given visual analog scale to record their pain p during the first week after each archwire placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for fixed appliance orthodontic treatment with 5-9 mm crowding of mandibular anterior teeth according to Little's irregularity index (LII).
2. Presence of all the mandibular permanent teeth, except the third molars.
3. Overbite and overjet that do not interfere with bracket placement on mandibular anterior teeth.
4. No history of trauma or root resorption in the mandibular incisors.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Less than 5 mm of mandibular incisors crowding (LII).
3. Severe crowding which requires treatment by extraction of premolars in the mandibular arch.
4. Blocked-out teeth that cannot be engaged with the aligning archwire.
5. Prior experience of periodontal disease and loss of attachment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Changes in alignment of anterior teeth will be measured using Little's irregularity index | 16 weeks
  A good-quality alginate impression for the lower arch should be taken pre-treatment and after 4, 8, 12 and 16 weeks and a stone study model is obtained. This study model which should be free from any discrepancy (such as bubbles) will be used to measure Little's irregularity index using a digital Vernier caliper to calculate the amount of mesial and distal contact displacement from the mesial contact surface of right mandibular canine to that on the other side, to the nearest 0.01 mm. The sum of these measurements represents the amount of Little's irregularity index.

SECONDARY OUTCOMES:
Root resorption using the scoring index that was provided by Malmgren et al. (1982) | 16 weeks
  Root resorption will be evaluated for the mandibular central incisors using periapical radiographs with digital sensors, and the worst score for either left or right central will be taken using the scoring index by Malmgren et al. (1982):
  * Grade 1: Irregular apical root contour.
  * Grade 2: Minor apical root resorption, a small area of root loss amounting to less than 2 mm.
  * Grade 3: Severe apical root resorption from 2 mm to one third of the original root length.
  * Grade 4: Extreme apical root resorption exceeding one third of the original root length.
pain perception using visual analog scale | 1st week after each wire placement.
  Evaluations of pain/discomfort will be made in the evening on a daily basis over the first seven days after bonding using a 10-point visual analog scale (VAS) with 0 refers to "no pain" and 10 refers to "intolerable pain". The participants will be reminded daily by a phone call or a text message to mark the recording sheet and will be asked to bring it on their next appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Yassir A. Yassir, M.Sc., P.hd. (UK), Study Director — University of Baghdad
Locations (1):
- Baghdad college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atik E, Gorucu-Coskuner H, Akarsu-Guven B, Taner T. A comparative assessment of clinical efficiency between premium heat-activated copper nickel-titanium and superelastic nickel-titanium archwires during initial orthodontic alignment in adolescents: a randomized clinical trial. Prog Orthod. 2019 Dec 16;20(1):46. doi: 10.1186/s40510-019-0299-4. PMID 31840204
- [Background] Azizi F, Extiari A, Imani MM. Tooth alignment and pain experience with A-NiTi versus Cu-NiTi: a randomized clinical trial. BMC Oral Health. 2021 Sep 6;21(1):431. doi: 10.1186/s12903-021-01789-5. PMID 34488744
- [Background] Berger J, Waram T. Force levels of nickel titanium initial archwires. J Clin Orthod. 2007 May;41(5):286-92. No abstract available. PMID 17652862
- [Background] Fleming PS, Johal A. Self-ligating brackets in orthodontics. A systematic review. Angle Orthod. 2010 May;80(3):575-84. doi: 10.2319/081009-454.1. PMID 20050755
- [Background] Gil FJ, Planell JA. Effect of copper addition on the superelastic behavior of Ni-Ti shape memory alloys for orthodontic applications. J Biomed Mater Res. 1999;48(5):682-8. doi: 10.1002/(sici)1097-4636(1999)48:53.0.co;2-m. PMID 10490682
- [Background] Jian F, Lai W, Furness S, McIntyre GT, Millett DT, Hickman J, Wang Y. Initial arch wires for tooth alignment during orthodontic treatment with fixed appliances. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD007859. doi: 10.1002/14651858.CD007859.pub3. PMID 23633347
- [Background] Kapila S, Sachdeva R. Mechanical properties and clinical applications of orthodontic wires. Am J Orthod Dentofacial Orthop. 1989 Aug;96(2):100-9. doi: 10.1016/0889-5406(89)90251-5. PMID 2667330
- [Background] Mahmoudzadeh M, Farhadian M, Alijani S, Azizi F. Clinical comparison of two initial arch wires (A-NiTi and Heat Activated NiTi) for amount of tooth alignment and perception of pain: A randomized clinical trial. Int Orthod. 2018 Mar;16(1):60-72. doi: 10.1016/j.ortho.2018.01.007. Epub 2018 Feb 23. PMID 29478933
- [Background] Montasser MA, Keilig L, Bourauel C. Archwire diameter effect on tooth alignment with different bracket-archwire combinations. Am J Orthod Dentofacial Orthop. 2016 Jan;149(1):76-83. doi: 10.1016/j.ajodo.2015.06.026. PMID 26718381
- [Background] Nabbat SA, Yassir YA. A clinical comparison of the effectiveness of two types of orthodontic aligning archwire materials: a multicentre randomized clinical trial. Eur J Orthod. 2020 Dec 2;42(6):626-634. doi: 10.1093/ejo/cjz102. PMID 32011678
- [Background] Papageorgiou SN, Konstantinidis I, Papadopoulou K, Jager A, Bourauel C. A systematic review and meta-analysis of experimental clinical evidence on initial aligning archwires and archwire sequences. Orthod Craniofac Res. 2014 Nov;17(4):197-215. doi: 10.1111/ocr.12048. Epub 2014 May 29. PMID 24889143
- [Background] Rucker BK, Kusy RP. Theoretical investigation of elastic flexural properties for multistranded orthodontic archwires. J Biomed Mater Res. 2002 Dec 5;62(3):338-49. doi: 10.1002/jbm.10325. PMID 12209919
- [Background] Sebastian B. Alignment efficiency of superelastic coaxial nickel-titanium vs superelastic single-stranded nickel-titanium in relieving mandibular anterior crowding: a randomized controlled prospective study. Angle Orthod. 2012 Jul;82(4):703-8. doi: 10.2319/072111-460.1. Epub 2011 Oct 19. PMID 22011096
- [Background] Wang Y, Liu C, Jian F, McIntyre GT, Millett DT, Hickman J, Lai W. Initial arch wires used in orthodontic treatment with fixed appliances. Cochrane Database Syst Rev. 2018 Jul 31;7(7):CD007859. doi: 10.1002/14651858.CD007859.pub4. PMID 30064155
- [Background] Malmgren O, Goldson L, Hill C, Orwin A, Petrini L, Lundberg M. Root resorption after orthodontic treatment of traumatized teeth. Am J Orthod. 1982 Dec;82(6):487-91. doi: 10.1016/0002-9416(82)90317-7. PMID 6961819
- [Derived] Noori RM, Ahmed OK, Kadhum AS, Yassir YA, Di Blasio M, Russo D, Cicciu M, Minervini G. The Effectiveness of Conventional and Advanced Aligning Archwires: The Insights of Two Randomized Clinical Trials. Eur J Dent. 2025 Oct;19(4):985-997. doi: 10.1055/s-0044-1795080. Epub 2025 Apr 4. PMID 40185146
- [Derived] Noori RM, Yassir YA. Effectiveness of tubular coaxial nickel-titanium and copper nickel-titanium orthodontic aligning archwires: A randomized clinical trial. Int Orthod. 2023 Dec;21(4):100812. doi: 10.1016/j.ortho.2023.100812. Epub 2023 Sep 28. PMID 37776695

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05391542/Prot_SAP_ICF_000.pdf